CLINICAL TRIAL: NCT06384729
Title: Effectiveness of the EXOPULSE Mollii Ⓡ Suit in Patients With Multiple Sclerosis: Randomized Clinical Trial
Brief Title: Effectiveness of the EXOPULSE Mollii Ⓡ Suit in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2024-04-08; First posted 2024-04-25 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: A randomized, double-blind clinical trial is proposed, in which two researchers will conduct the intervention, and a third researcher will be responsible for programming the suits and attaching the belt to the suit. The data will be analyzed by a fourth researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exopulse on group (Experimental): An individual assessment will be conducted to determine the parameters of the suit, and they will wear the suit for 60 minutes three times a week for three weeks. An initial assessment will be conducted, followed by another assessment after the 3-week treatment period.
  Interventions: Device: EXOPULSE Mollii Ⓡ
- Exopulse of group (Placebo Comparator): The suit will be worn with the parameters set to 0 for 60 minutes, three times a week, for three weeks. An initial assessment will be conducted, followed by another assessment after the 3-week treatment period.
  The suit will be worn with the parameters set to 0 for 60 minutes, three times a week, for three weeks. An initial assessment will be conducted, followed by another assessment after the 3-week treatment period.
  Interventions: Device: EXOPULSE Mollii Ⓡ

INTERVENTIONS:
Device: EXOPULSE Mollii Ⓡ — The EXOPULSE Mollii method (EXONEURAL NETWORK AB, Danderyd, Sweden) is an innovative approach to non-invasive and self-administered electrical stimulation with multiple electrodes incorporated into a full-body suit. It consists of comfortable, breathable, and washable synthetic material pants and a jacket. It has been primarily designed to reduce disabling spasticity and improve motor function. The method refers to the concept of reciprocal inhibition induced by stimulating the antagonist of a spastic muscle, at low frequencies and intensities, which is considered to reduce spasticity.

SUMMARY:
Abstract:

Background:

Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the central nervous system with unknown etiology, causing a variety of symptoms including impaired balance, coordination, and walking difficulties. The Exopulse Mollii Ⓡ suit is an innovative approach for non-invasive, self-administered electrical stimulation designed to alleviate spasticity and improve motor function in various neurological conditions.

Objective:

To determine the effectiveness of the Exopulse Mollii Ⓡ suit in improving motor control in patients with MS.

Methods:

A randomized, double-blind clinical trial will be conducted, recruiting patients diagnosed with MS , aged 18 or above, with a Functional Ambulation Category (FAC) score between 2 and 4. Patients will be randomly assigned to two groups receiving either inactive or active Exopulse Mollii Ⓡ treatment for 60 minutes, three times a week, for three weeks. Outcome measures include pain, balance, gait speed, risk of falls, perception of walking difficulties, and quality of life assessed using validated scales. Statistical analysis will be performed using SPSS v.29.0.0.0.

Results:

Data on age, sex, weight, and MS-related factors will be collected at baseline. Primary outcomes include changes in pain, balance, and gait speed, while secondary outcomes encompass risk of falls, perception of walking difficulties, and quality of life. Analysis will compare mean differences between groups using appropriate statistical tests.

Conclusion:

This study aims to evaluate the efficacy of the Exopulse Mollii Ⓡ suit in enhancing motor function in MS patients. Findings may contribute to the development of novel therapeutic strategies for managing MS-related symptoms and improving patients' quality of life.

DETAILED DESCRIPTION:
Introduction:

Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the central nervous system with unknown etiology. Common symptoms include fatigue, visual disturbances, balance and coordination problems, sensory disturbances, spasticity, cognitive and emotional disorders, speech impairments, bladder and bowel issues, and sexual dysfunction. MS affects approximately 2.2 million people worldwide. Gait abnormalities are a distinctive feature of MS and a significant cause of disability and reduced health-related quality of life. Individuals with MS typically exhibit slower walking speeds, lower cadence, and increased variability between strides, attributed to demyelination resulting in reduced conductivity in the somatosensory nervous system, decreased muscle strength, vestibular dysfunction, and severe fatigue.

The EXOPULSE Mollii Ⓡ method is an innovative approach to non-invasive, self-administered electrical stimulation using multiple electrodes incorporated into a full-body suit. Comprising comfortable, breathable, and washable synthetic material, the Mollii Ⓡ suit primarily aims to alleviate disabling spasticity and enhance motor function. The method operates on the concept of reciprocal inhibition induced by stimulating the antagonist of a spastic muscle at low frequencies and intensities, thus considered to reduce spasticity. Moreover, the EXOPULSE Mollii Ⓡ suit has demonstrated benefits in children with cerebral palsy, spasticity, and chronic stroke patients. Therefore, this study aims to evaluate the effects of a 60-minute session with the EXOPULSE Mollii Ⓡ suit on patients with multiple sclerosis.

Methodology:

A randomized, double-blind clinical trial will be conducted, with two investigators performing the intervention and a third responsible for programming the suits and attaching the belt. Patients will be recruited from the Fivan Foundation, where the intervention will take place. Recruitment and patient selection will be conducted through therapists at the center, informed in advance about the project's content. The suits, provided by the Fivan Foundation and Ottobock, consist of comfortable, breathable, and washable synthetic pants and jackets. Patients meeting the following inclusion criteria will be selected:

* Diagnosed with multiple sclerosis by their physician
* Aged 18 or above.
* Able to understand verbal commands.
* Having a Functional Ambulation Category (FAC) score between 2 and 4.

Exclusion criteria include:

* Pregnancy.
* Having an intrathecal baclofen pump.
* Having received botulinum toxin infiltration in the last 3 months.
* Wearing electronic or magnetic medical devices (pacemakers, shunts, etc.) that may be affected by magnets.
* BMI > 35.

Patients will be randomly divided into two groups using a coin toss method. An initial individual assessment session will be conducted, including randomization, providing each patient with an assessment sheet, and obtaining informed consent. The control group will wear the Exopulse Mollii Ⓡ suit with parameters set to 0, while the second group will wear the same suit with parameters adjusted to each individual assessment. Both groups will undergo 60-minute sessions, three times a week for three weeks, to assess potential beneficial effects of this device for MS patients. At three weeks, a crossover will occur, with the group initially having parameters set to 0 now receiving treatment for another 3 weeks, while the other group will have the treatment discontinued to assess maintenance of effects. Initial, 3-week, and 6-week assessments will be conducted for both groups using previously validated scales detailed in the following section. This intervention will be added to the patient's usual treatment without interfering with it. Sample size was determined using the GRANMO© program, with 11 subjects per group, considering an alpha risk of 0.05, a beta risk below 0.2 in a bilateral contrast, and an estimation based on a common standard deviation of 4.89, taking into account a 5% follow-up loss rate.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of Multiple Sclerosis as confirmed by a physician using McDonald's criteria.

  * Age over 18 years.
  * Ability to comprehend verbal commands.
  * Scoring between 2 and 4 on the Functional Ambulation Category (FAC).

Exclusion Criteria:

* Pregnancy.

  * Having an intrathecal baclofen pump.
  * Having received botulinum toxin injections in the last 3 months.
  * Wearing electronic or magnetic medical devices (pacemakers, shunts, etc.) that may be affected by magnets.
  * BMI > 35.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
referred pain | 3 weeks
  Visual analogue scale. Range: 0 to 10 Interpretation: Higher scores indicate higher levels of pain or symptoms.
Balance | 3 weeks
  Berg Balance Scale; Range: 0 to 56 Interpretation: Higher scores indicate better balance and motor function.
gait speed and distance | 3 weeks
  6 minutes walking test; Interpretation: Interpretation: Greater distances indicate better functional capacity and endurance.

SECONDARY OUTCOMES:
fall risk | 3 weeks
  Tinetti scale: Range: 0 to 28 Interpretation: Higher scores indicate better balance and mobility.
perception of walking difficulties | 3 weeks
  Multiple Sclerosis Walking Scale-12: Range: 0 to 100 Interpretation: Higher scores indicate greater difficulty walking and poorer mobility.
perceived quality of life | 3 weeks
  Multiple Sclerosis Impact Scale-29: Range: 29 to 116 Interpretation: Higher scores indicate greater impact on quality of life and higher disability due to multiple sclerosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Cecilia Estrada Barranco, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No